CLINICAL TRIAL: NCT07095413
Title: Assessing the Performance of Wesper Lab for Obstructive and Central Sleep Apnea Diagnosis in Adult Populations
Brief Title: Assessing the Performance of Wesper Lab for Obstructive and Central Sleep Apnea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wesper Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WSP-222
Record Dates: First submitted 2025-07-14; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive; Sleep Apnea, Central
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Intervention Model Description: All participants will wear the Wesper Lab sensors while undergoing the Polysomnography (PSG) test. The study focuses on evaluating the performance of the Wesper Lab sensors in the context of standard PSG without a separate control or comparison group.
Masking Description: A blinding model will be implemented for the scoring of the Wesper Lab data and Polysomnography (PSG) to minimize bias during the scoring and analysis of sleep study data.
  All sleep study recordings are disidentified before being presented to the readers. The primary reader and any additional secondary readers will be blinded to which device was used to collect the data (Wesper Lab vs. PSG). Studies will be reviewed in a predetermined randomized order to further prevent any bias. All data will be presented using the same viewing and scoring platform, ensuring consistency in how the data is labeled and displayed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medical Device: Wesper Lab Home Sleep Apnea Test (Other): This arm consists of participants who will undergo an overnight polysomnography (PSG) evaluation while simultaneously wearing the Wesper Lab home sleep apnea tests.
  Interventions: Diagnostic Test: Wesper Lab Home Sleep Apnea Test

INTERVENTIONS:
Diagnostic Test: Wesper Lab Home Sleep Apnea Test — Subjects will wear the Wesper Lab home sleep apnea tests, which includes 2 wireless sensors and a pulse oximeter.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the Wesper Lab home sleep apnea test as a tool to aid in the diagnosis of sleep apnea in adult patients (age ≥21 years) who are recommended for an overnight polysomnography (PSG) evaluation. The main questions it aims to answer are:

1. Is Wesper Lab home sleep apnea test as accurate as an in-laboratory sleep study (polysomnography) for the diagnosis of obstructive and central sleep apnea?
2. Is Wesper Lab accurate in a wide range of body types and skin types?

Participants will:

1. Provide informed consent and complete a brief medical history.
2. Undergo an overnight polysomnography sleep study while wearing two Wesper Lab patches and a compatible pulse oximeter.
3. Have a follow-up communication within 5 days post-study to assess any adverse events.

DETAILED DESCRIPTION:
This study aims to validate the Wesper Lab wireless sensors as a reliable alternative to traditional PSG for diagnosing sleep apnea, potentially providing a more convenient method for patients while maintaining diagnostic accuracy. The structured approach to data collection, monitoring, and follow-up underscores a thorough methodology to assess both effectiveness and safety. The study is a single-center, single-arm clinical trial designed to evaluate the effectiveness of the Wesper Lab wireless sensors for aiding in the diagnosis of sleep apnea, specifically comparing its performance to overnight polysomnography (PSG).

The primary aim is to determine how well the Wesper Lab wireless sensors correlate with traditional PSG results in measuring obstructive sleep apnea (OSA) and central sleep apnea (CSA) through key metrics, specifically the apnea-hypopnea index (AHI) and central apnea/hypopnea index (CAHI).

Approximately 100 eligible adult patients (≥21 years) who have been referred by a physician for an overnight PSG test to evaluate sleep apnea.

Patients will undergo PSG testing while simultaneously wearing two Wesper Lab sensors and a compatible pulse oximeter for one night at the clinic. Sleep technicians will monitor and set up the devices, and data will be collected via a smartphone app linked to the Wesper Lab system. The PSG will record brain activity, blood oxygen levels, heart rate, breathing patterns, and movements. Data will be collected during the sleep period, and post-study, the signals will be analyzed by qualified readers who are blinded to the device used for data collection.

To demonstrate that the correlation between the AHI/CAHI from the Wesper Lab and PSG exceeds a predefined performance goal (PG) using Pearson correlation. To establish that the 95% limits of agreement between AHI/CAI from the two devices fall within acceptable upper and lower limits. Evaluate inter-rater reliability of AHI/CAHI readings. Assess agreement in apnea classification (mild, moderate, severe) between the two methods.

Analyze differences based on sleep position (supine vs. non-supine).

The primary safety endpoints include tracking adverse events (AEs) and serious adverse events (SAEs) related to the use of the Wesper Lab device throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age
* Have a referral to the study site from a physician to complete an overnight polysomnogram test for sleep apnea detection or follow-up.
* Be willing and able to wear two Wesper Lab patches and an FDA-cleared pulse oximeter in conjunction with a polysomnogram, for a single night.
* Be able and voluntarily willing to sign a written informed consent form prior to the initiation of any study procedures. Adult patients unable to provide written informed consent on their own behalf will not be eligible for the study.

Exclusion Criteria:

* Women who are pregnant, trying to get pregnant or who have a positive urine pregnancy test on the day of the study.
* Women who are breast-feeding
* History of severe insomnia
* Any known health condition that, in the opinion of the Investigator, would exclude the patient from participating in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of the Apnea/Hypopnea Index Between Wesper Lab Sensors and PSG | 8 Hours
  The primary outcome measure is to assess the correlation between the apnea-hypopnea index (AHI) and obtained from the Wesper Lab wireless sensors and those derived from the polysomnography (PSG) recordings.
Correlation of the Central Apnea/Hypopnea Index Between Wesper Lab Sensors and PSG | 8 Hours
  The primary outcome measure is to assess the correlation between the apnea-hypopnea index (CAHI) and obtained from the Wesper Lab wireless sensors and those derived from the polysomnography (PSG) recordings.

SECONDARY OUTCOMES:
Inter-Rater Reliability | 8 Hours
  Assess the consistency of signal scoring among different readers using the Wesper Lab device.
Agreement in Apnea Classification | 8 Hours
  Evaluate the concordance between the Wesper Lab sensors and PSG in classifying the severity of apnea (mild, moderate, severe).
Classification of Apnea Type | 8 hours
  To determine the agreement between the Wesper Lab sensors and PSG in identifying the type of apnea (Obstructive Sleep Apnea (OSA) vs. Central Sleep Apnea (CSA)).
Agreement in Respiratory Event Detection by Optical Sensors - AHI | 8 Hours
  To determine the agreement between the Wesper Lab optical sensors and PSG in determining the apnea/hypopnea index (AHI).
Agreement in Total Sleep Time by Optical Sensors | 8 Hours
  To determine the agreement between the Wesper Lab optical sensors and PSG for estimating total sleep time.
Agreement in Respiratory Event Detection by Optical Sensors - CAHI | 8 Hours
  To determine the agreement between the Wesper Lab optical sensors and PSG in determining the central apnea/hypopnea index (CAHI).

CONTACTS AND LOCATIONS:
Overall Officials: Chelsie E Rohrscheib, Ph.D, Study Director — Attend a workshop; Ruchir P Patel, M.D., Principal Investigator — The Insomnia and Sleep Institute of Arizona

IPD SHARING:
Plan to Share IPD: No
No IPD will be available to share with researchers no associated with Wesper Inc.